CLINICAL TRIAL: NCT06572475
Title: USPIO Enhanced MR Imaging in CNS Tumours (UMIC) : A Pilot Study of Ferumoxytol (Feraheme ©) as an Imaging Biomarker of Tumour Associated Macrophage (TAM) Infiltration in Vestibular Schwannoma (VS) and Transforming Low Grade Glioma (LGG)
Brief Title: USPIO Enhanced MR Imaging in CNS Tumours (UMIC)
Acronym: UMIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22NEURO06-S
Record Dates: First submitted 2024-06-15; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Vestibular Schwannoma; Glioma, Astrocytic
MeSH Terms: conditions — Neuroma, Acoustic; Astrocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trial arm 1 (Experimental): Group A: Patients with sporadic VS undergoing radiological surveillance (n=12). The sample will include growing tumours (n=6) that are being considered for surgical resection, and non-growing/static tumours (n=6) that are being considered for either further radiological surveillance or surgery.
  Group B: Patients with suspected transforming low-grade glioma (n=5). Patients in this cohort will have a proven or suspected diagnosis of low-grade glioma (LGG) but with features on routine clinical imaging suggestive of malignant transformation to either grade III (anaplastic) or grade IV glioma. Patients with suspected transforming LGG who are listed to undergo surgical resection will be enrolled into the study so that acquired imaging can be compared with tissue datasets.
  Interventions: Diagnostic Test: USPIO enhanced MRI

INTERVENTIONS:
Diagnostic Test: USPIO enhanced MRI — Ferumoxytol (Feraheme©, AMAG pharmaceuticals, US) enhanced MRI

SUMMARY:
The immune response or inflammation is known to be a key driver of progression and growth in many solid tumours. Inflammatory cells called macrophages are present in high numbers in many brain tumours and these tumour associated macrophages or TAM are thought to have prognosis and treatment implications in these tumours. A key question, however, is how this inflammation or TAM abundance can be detected, measured and monitored in the clinic. A clinically applicable imaging test that can directly and accurately measure tumour macrophage content would be of considerable value and one technique that may provide this is USPIO enhanced magnetic resonance imaging (MRI). Following intravenous injection, USPIO or ultrasmall superparamagnetic iron oxide nanoparticles, circulate in the bloodstream before being taken up by inflammatory cells/macrophages in tumour tissue, wherein they can be detected by MRI. This pilot study is to evaluate if a commercially available USPIO preparation called ferumoxytol (Feraheme ©) can accurately quantify macrophage abundance in brain tumours, with an exploratory focus on vestibular schwannoma (VS) and suspected transforming low-grade glioma (LGG). Patients with both non-growing (static) and growing VS, and patients with suspected transforming LGG will undergo dedicated MRI sequences before, immediately after (< 2 hours) and at both 24 and 48hrs after ferumoxytol administration. In patients undergoing surgery, acquired imaging will be compared with resected tumour tissue so that markers of inflammation can be compared with USPIO uptake. Through advanced laboratory methods this study will seek to establish within resected VS and LGG specimens: the cellular destination/s of USPIO uptake; the nature of the inflammatory and/or tumour cells containing the USPIO; and the relationship between USPIO uptake and tumour blood vessel permeability or leakiness.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 16 years old
* Have a CNS tumour suspected to be one of the defined histological types (vestibular scwhannoma or low grade glioma)
* Be able to lie still for up to 1 hour comfortably
* Opinion of the treating clinician is that the patient will be able to successfully complete the research imaging protocol.

Exclusion Criteria:

* Life expectancy less than 1 year
* Previous CNS radiotherapy/ stereotactic radiosurgery (SRS)
* Females who are pregnant/ breastfeeding
* Patients with an eGFR < 30ml/min
* Patients with known and documented history of iron overload/haemosiderosis/ haemochromatosis
* Patients with immune or inflammatory conditions e.g. systemic lupus erythematous, rheumatoid arthritis
* Patients with absolute (e.g. pacemaker) and relative (anxiety or claustrophobia) contraindications to MR scanning
* Patients with a history of allergic reaction to iron or dextran
* Patients with a history of allergic reaction to gadolinium contrast agents, asthma or renal problems
* Patients who are unable to adequately understand verbal explanations or written information given in English.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Establish in a cohort of surgically resected sporadic VS if the enhancement pattern of delayed (24-48 hr) USPIO uptake correlates with tissue markers of TAM density and tissue microvascular markers. | Three years
  Use correlation tests to establish the relationship between delayed (24-48 hr) USPIO related MRI signal intensity changes and tissue markers of TAM density and microvascular markers.
Establish the relationship between enhancement patterns following GBCA administration and the volume, pattern and intensity of early (<2hr) and delayed (24-48 hr) USPIO imaging in these tumours. | Three years
  Differences in the enhancement pattern between post GBCA T1W images and the delayed (24-48hr) ferumoxytol enhanced T1W images will be compared through visual inspection and use of the structural similarity index
Evaluate the association between microvascular parameters derived from dynamic contrast enhanced (DCE) MRI) and the volume, pattern and intensity of early (<2hr) and delayed (24-48 hr) USPIO imaging in these tumours. | Three years
  Use voxelwise correlation tests and ROI analysis to establish the relationship between microvascular parameters derived from dynamic contrast enhanced (DCE) MRI) and USPIO related signal intensity changes at early (<2hr) and delayed (24-48 hr) imaging timepoints in these tumours.
Establish in VS the relationship between the volume, pattern and intensity of early (<2hr) and delayed (24-48 hr) USPIO imaging in these tumours with tumour size and tumour growth status (non-growing or static vs growing). | Three years
  Evaluate using appropriate parametric and non-parametric statistical tests if there are differences between non-growing and growing VS in USPIO related signal intensity changes on acquired T1, T2 and T2* weighted imaging at early (<2hr) and delayed (24-48 hr) imaging timepoints. Evaluate using correlation and regression analyses if there is a relationship between tumour size and USPIO related signal intensity changes on acquired T1, T2 and T2* weighted imaging at early (<2hr) and delayed (24-48 hr) imaging timepoints.
Establish within resected VS and transforming low-grade glioma specimens the cellular destination/s of USPIO internalisation and the in vivo relationship between BBB disruption and USPIO extravasation. | Three years
  Immunohistochemistry (IHC)/ immunofluorescence will be used on both formalin fixed paraffin embedded (FFPE) and frozen tissue samples to map the uptake of USPIO within immune and non-immune cell populations.
Establish if the enhancement pattern of delayed (24-48 hr) USPIO uptake correlates with loco-regional tissue markers of immune cell infiltration and malignant transformation within imaged transforming low grade glioma. | Three years
  Evaluate using appropriate parametric and non-parametric statistical tests if there are differences in USPIO related signal intensity changes and immune cell infiltration within regions of histologically proven transformation when compared to non-transformed areas.

CONTACTS AND LOCATIONS:
Overall Officials: David Coope, PhD FRCS(SN), Principal Investigator — Northern Care Alliance NHS Foundation Trust
Locations (1):
- Salford Royal Hospital Northern Care Alliance NHS Foundation Trust, Salford, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No